CLINICAL TRIAL: NCT04167007
Title: Randomized Phase 3 Trial Comparing FOLFOX to Gemcitabine in Metastatic First-line in Patients With Pancreatic Adenocarcinoma and Non-fit for FOLFIRINOX
Brief Title: FOLFOX vs Gemcitabine in Patients With Metastatic Pancreatic Cancer Non-fit to FOLFIRINOX
Acronym: GEMFOX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D20180177; 2019-001364-30 (EudraCT Number)
Record Dates: First submitted 2019-08-28; First posted 2019-11-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; Metastasis; Gemcitabine; FOLFOX; first-line
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Gemcitabine; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Gemcitabine at 1000 mg/m²
  Interventions: Drug: Gemcitabine
- Group II (Active Comparator): Oxaliplatin at 85 mg/m² ; Folinic acid 400 mg/m² (racemic form) or 200 mg/m² (L-form) and 5-FU 2400 mg/m²
  Interventions: Drug: FOLFOX

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine at 1000 mg/m² as intravenous (IV) infusion over 30-40 minutes on days 1, 8, and 15, followed by 1 week of rest, every 28 days
  Arms: Group I
Drug: FOLFOX — Oxaliplatin at 85 mg/m² given as a 2 hours IV infusion on days 1 and 15; Folinic acid 400 mg/m² (racemic form) or 200 mg/m² (L-form) in 250 ml glucose 5% solution given as a 2 hours IV infusion on days 1 and 15; and 5-FU 2400 mg/m² administered as continuous 46-hour IV infusion on days 1-3 and 15-17, every 28 days.
  Arms: Group II

SUMMARY:
Pancreatic adenocarcinoma (PAC) incidence increases regularly in Western countries and it is expected to become the second leading cause of cancer-related mortality in 2020. The prognosis of this disease remains very poor with an overall 5-year survival rate less than 5%.

The FOLFIRINOX regimen (5-fluorouracil [5-FU], folinic acid, irinotecan, and oxaliplatin) and the combination of nab-paclitaxel with gemcitabine demonstrated to be more effective than gemcitabine alone, and are both validated as standard first-line treatment options for metastatic PAC. However, the use of FOLFIRINOX is limited to patients with ECOG performance status (PS) 0-1 and aged less than 75 years. Nab-paclitaxel is currently not reimbursed in France.

DETAILED DESCRIPTION:
This trial is an open label, multicenter, randomized phase III trial comparing gemcitabine vs FOLFOX in patients with metastatic pancreatic adenocarcinoma and non-fit for FOLFIRINOX. Adults fulfilling inclusion criteria and non-inclusion criteria will be randomized between a FOLFOX arm and a gemcitabine arm. The primary endpoint is the overall survival (OS) at 24 months. The secondary objectives are : objective response rate and disease control rate (RECIST v1.1, in case of evaluable lesion), duration of response, duration of disease control, progression free survival (PFS), the evolution of biomarkers Ca 19-9 and CEA under treatment, the toxicities according to International Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, the safety of both arms, the quality of life, the dose intensity (DI) of each protocol, the Quality-Adjusted Survival, and the rate and type of second-line / third-line regimens chemotherapy. With an expected median survival time in the control group of 5 months, an accrual period of 3 years and a minimum follow-up period of 2 years, a total of 199 patients per group are required to detect a hazard ratio of 0.75 based on a 5% two-sided type I error rate and a power of 80%, leading to a total number of 400 patients to include.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically or cytologically proven adenocarcinoma of the pancreas,
3. In absence of histologically or cytologically proven adenocarcinoma, a cluster of clinical, biological and radiological arguments consistent with the diagnosis: among these, a hypodense pancreatic tumor at CT and a Ca 19-9 greater than 500 UI/ml are essential prerequisites,
4. Metastatic disease confirmed (stage IV),
5. No prior therapy for metastatic disease (in case of previous adjuvant therapy, interval from end of chemotherapy and relapse must be >12 months),
6. Age ≥18 years ,
7. Patient non-fit for FOLFIRINOX,
8. For patients with ECOG performance status (PS ) ≥2, an albuminemia level >25 g/l is required,
9. Haematological status: neutrophils (ANC) >2x109/L; platelets >100x109/L; haemoglobin ≥9g/dL,
10. Adequate renal function: serum creatinine level <150μM, and estimated creatinine clearance >30ml/min,
11. Adequate liver function: AST (SGOT) and ALT (SGPT) ≤2.5xULN (≤5xULN in case of liver metastases),
12. Total bilirubin ≤3 x ULN,
13. QT / QTc interval at baseline ECG (performed within 1 month before randomization) < than 450 msec for men and < than 470 msec for women,
14. Baseline evaluations performed before randomization: clinical and blood evaluations no more than 2 weeks (14 days) prior to randomization, tumor assessment (CT-scan or MRI, evaluation of non-measurable lesions) no more than 3 weeks (21 days) prior to randomization,
15. Female patients must be surgically sterile, or be postmenopausal, or must commit to using reliable and appropriate methods of contraception during the study and during at least six months after the end of study treatment (when applicable). All female patients with reproductive potential must have a negative pregnancy test (β HCG) within 7 days prior to starting protocol treatment. Breastfeeding is not allowed.
16. Male patients must agree to use effective contraception in addition to having their partner use a contraceptive method as well during the trial and during at least six months after the end of the study treatment
17. Affiliation to a French social security system (recipient or assign).

Exclusion Criteria:

1. History or evidence upon physical examination of CNS metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy),
2. Local or locally advanced disease (stage I to III),
3. Patient uses warfarin,
4. Patient receiving concomitant radiotherapy,
5. Electrolytic report uncontrolled: hypercalcemia and/or hypokalemia and/or hypomagnesemia,
6. Pre-existing permanent neuropathy (NCI grade ≥2 ),
7. Poor nutritional status
8. Known dihydropyrimidine dehydrogenase (DPD) total or partial deficiency (DPD activity dosage at inclusion visit),
9. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy),
10. Treatment with any other investigational medicinal product within 28 days prior to study entry,
11. Other serious and uncontrolled non-malignant disease (eg. active infection requiring systemic therapy, coronary stenting or myocardial infarction or stroke in the past 6 months),
12. Known or historical active infection with HIV, or known active infection untreated with hepatitis B or hepatitis C ,
13. Known uncontrolled bacterial infection
14. History or active interstitial lung disease (ILD),
15. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
16. Patients with known allergy to active substance or any excipient of study drugs,
17. Allergy to iodinated contrast product
18. Concomitant administration of live, attenuated virus vaccine and concomitant administration of prophylactic phenytoin.
19. Patients under legal protection or unable to consent
20. Participation in another interventional research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) at 24 months | At 24 months after inclusion
  OS will be defined as the delay between the date of inclusion and the date of death (whatever the cause) or the date of last news if the patient is alive.

SECONDARY OUTCOMES:
Objective response rate | At 24 months after inclusion
  RECIST criteria 1.1 in case of evaluable lesion
Disease control rate | At 24 months after inclusion
  RECIST criteria 1.1 in case of evaluable lesion
Duration of response | Tumor assessment will be done every 2 cycles (1cycle = 28 days), assessed up to 24 months after inclusion
  The time interval between the first occurrence of partial or complete response according to RECIST criteria and secondary progression (clinic or radiologic)
Duration of disease control | Tumor assessment will be done every 2 cycles (1 cycle = 28 days), assessed up to 24 months after inclusion
  The time interval between the first occurrence of disease control (stabilization or partial response or complete response) according to RECIST criteria and secondary progression (clinic or radiologic)
Progression Free Survival (PFS) | From inclusion to the date of first event (progression or death) or date of last news if the patient is alive without progression, assessed up to 60 months
  In most cases, patient will have a radiologic evaluation and radiologic progression will be defined according to RECIST criteria. In absence of radiologic evaluation (decision of investigator), clinic progression would be defined by investigators according to clinical deterioration of PS, increase of symptoms, and/or increase of tumor markers.
Carbohydrate antigen 19-9 (CA-19-9) and carcinoembryonic antigen (CEA) levels | At baseline (at selection or inclusion visit before starting treatment) and then each 2 cycles (every 8 weeks) until end of treatment, up to 24 months
Toxicities: Type, frequency and severity of adverse events and serious adverse events | From inclusion to end of treatment, up to 24 months
  Toxicities will be described and grades according to International Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Safety: Rate of serious adverse events, grade 3-4 toxicities (hematologic and non-hematologic) | From inclusion to end of treatment, up to 24 months
  Rate of serious adverse events, grade 3-4 toxicities (hematologic and non-hematologic). Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
inLongitudinal changes in Quality of life (EORTC QLQ C-30 questionnaire and a consensual geriatric minimum data set (SOFOG) for patients ≥75 years) | At inclusion, before starting treatment, and then Day 1 of each cycle (every 4 weeks, 1 cycle = 28 days) until end of treatment, up to 24 months
  Quality of life will be studied by means of the EORTC QLQ C-30 questionnaire (30 questions, score from 30 to 126) and a consensual geriatric minimum data set (SOFOG: 7 questions, score from 0 to 24) for patients ≥75 years at inclusion and at each cycle. A 5-point deterioration in HRQoL scores will be considered as the minimal clinically important difference (MCID). Time until MCID will be analyzed (for each questionnaire) and compared between the two groups. The dynamic change under treatment will be compared at each cycle.
Dose intensity of each protocol | During the entire treatment period, up to 24 months
  The dose intensity (DI) of each protocol will be calculated based on the number of cycles received by each patient. The relative DI will be calculated as the ratio of the DI to the DI indicated in the protocol (obtained as the dose specified per cycle in mg/m²)
Quality-adjust Time Without Symptoms of disease or Toxicities (Q-TWiST) | During the entire treatment period, up to 24 months
  The Q-TWiST method combines treatment benefits and risks into a single measure by partitioning survival time into three health states and subsequently assigning quality-of life weights to the survival time in each state. The primary Q-TWiST analysis will be performed using the Intention-to-treat analysis(ITT) population, and will be supplemented with analyses in the per-protocol population (i.e., patients who received ≥80% of the protocol-defined treatment during the first 6 weeks of treatment) and analysed in pre-specified subgroups: age (<75 years, ≥75 years), baseline PS (0-1, 2), liver metastases (Yes, No), and tumour location (head, other).
Rate of second and third line | From end of study treatment to patient death, assessed up to 60 months.
  For the patients who will stop the treatment of the protocol (for progression, toxicity or other reason...), we will register the date of beginning and of last administration of each new line of chemotherapy administered during the follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste BACHET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- APHP - Groupe Hospitalier Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No